CLINICAL TRIAL: NCT05582733
Title: Effects of Cervical Spine Manipulation on Upper Trapezius Active Versus Conventional Techniques.
Brief Title: Effects of Cervical Spine Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Collaborators: Riphah International University (Other)
Responsible Party: Principal Investigator, Madeeha Shafiq, Lecturer, University of Lahore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REC:00570
Record Dates: First submitted 2022-10-03; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Cervical Pain
MeSH Terms: conditions — Neck Pain | interventions — Traction

STUDY DESIGN:
Intervention Model Description: Control was treated with Manual Pressure release followed by stretching while in experimental received cervical spine manipulation (chin hold) kaltenborn followed by stretching.
Who Masked: Participant
Masking Description: Free envelop method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical spine manipulation (Experimental): In spinal manipulation, the velocity, magnitude and direction of the impulse are controlled to encourage relaxation and comfort of muscle and connective tissue.
  Interventions: Other: Cervical spine manipulation; Other: traction
- traction (Experimental): aimed to relieve pressure on the spine
  Interventions: Other: Cervical spine manipulation; Other: traction

INTERVENTIONS:
Other: Cervical spine manipulation — hot pack for 10 minutes will be applied followed by cervical manipulation (chin hold kaltenborn) once and then stretching
Other: traction — Hot pack will be applied followed by sustained pressure or MPR for 90 sec and then stretching.

SUMMARY:
To determine the immediate effects of cervical spine manipulation on pressure pain sensitivity on upper trapezius trigger point. it was a randomized control trial including 66 patients at physiotherapy OPD of railway rehabilitation center from August 2019 to December 2019, Railway General Hospital Pakistan and Max Rehab and decompression center Max health Hospital G8 Islamabad. The subjects were randomly divided into two groups (group control and experimental) by free envelope method.

DETAILED DESCRIPTION:
To determine the immediate effects of cervical spine manipulation on pressure pain sensitivity on upper trapezius trigger point and neck ranges of motion. A randomized control trial of 66 patients was conducted from August 2019 to December 2019 at physiotherapy OPD of railway rehabilitation center, Railway General Hospital Pakistan and Max Rehab and decompression center Maxhealth Hospital G8 Islamabad. The subjects were randomly divided into two groups (group control and experimental) by free envelope method. Control was treated with Manual Pressure release followed by stretching while in experimental received cervical spine manipulation (chin hold) kaltenborn followed by stretching. Structural questionnaire was used for pre and post assessment. Outcomes were measured by algometry and inclinometer before and after the application of respective techniques. The data was analyzed at baseline and immediately after the intervention on IBM SPSS-21.

ELIGIBILITY:
Inclusion Criteria:

* 1.presence MTrps in upper trapezius
* limited side bending and rotation
* both gender
* age between 25 to 45

Exclusion Criteria:

* Malignancy, infection, trauma, bone deformities.
* Acute Disc Protrusion
* Positive VBI
* Positive Sharp purser test
* History of whiplash injury

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
changes from the baseline in Algometer values | Baseline and 3 weeks
  It is a device used to identify the pressure and force eliciting a pressure pain threshold. The hand held algometer 1 cm round rubber surface which applies force and display for readings in newtons or kilograms.Sustained force is usually applied at the right angle to the soft tissue. Estimated pressure application rates have ranged from 0.05 to 20N/s. it has a high validity and reliability for measuring pain pressure threshold in patients of myofascial trigger points.
changes from the baseline in Inclinometer values | Baseline and 3 weeks
  It is a device used to measure neck ranges of motion.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, PHD*, Principal Investigator — ghafoor.sajjad@riphah.edu.pk
Locations (1):
- Dr. Abdul Gaffoor, Islamabad, Pakistan